CLINICAL TRIAL: NCT05519228
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the ToggleLoc™ 2.9mm Soft Tissue System (Implants and Instrumentation) in the Elbow - A Multicenter Retrospective Consecutive Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the ToggleLoc™ 2.9mm in the Elbow
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-72SM
Record Dates: First submitted 2022-06-01; First posted 2022-08-29 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2023-12

CONDITIONS: Epicondylitis of the Elbow; Biceps Tendon Disorder
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ToggleLoc 2.9 mm soft tissue device: Patients who already received the ToggleLoc 2.9 mm soft tissue device in the elbow. No additional surgery will be performed.
  Interventions: Device: ToggleLoc 2.9 mm Soft Tissue System

INTERVENTIONS:
Device: ToggleLoc 2.9 mm Soft Tissue System — The ToggleLoc 2.9 mm Soft Tissue System consist of non-resorbable device intended to aid in arthroscopic and orthopaedic reconstructive procedures requiring soft tissue to bone fixation

SUMMARY:
The study is a multicenter, retrospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to collect data confirming safety, performance and clinical benefits of the ToggleLoc 2.9 mm Soft Tissue System when used for soft tissue to bone fixation in the elbow. The primary objective is the assessment of performance by analyzing soft tissue to bone healing in the elbow.

The secondary objective is the assessment of safety and clinical benefits. Safety will be evaluated by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to device, instrumentation and/or procedure will be specified. Clinical benefits will be assessed by recording patient-reported outcome measures (PROMs) at the longest follow-up after surgery (minimum one year).

DETAILED DESCRIPTION:
The ToggleLoc 2.9 mm Soft Tissue System consist of non-resorbable device intended to aid in arthroscopic and orthopaedic reconstructive procedures requiring soft tissue to bone fixation. The clinical purpose is to restore the function and flexibility of the elbow requiring soft tissue to bone fixation and to relieve pain that cannot be controlled by other treatments.

Two sites will be involved in this study. The aim is to include a total of 83 consecutive series cases operated with the ToggleLoc 2.9 mm in the elbow. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop and intraop will be available in medical notes. The patients will be asked to complete patient questionnaires during a minimum 1 year follow up visit/phone call. In addition, any complications and adverse events that occured since the surgery will also be collected during the follow-up visit/phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received the ToggleLoc 2.9 mm Soft Tissue device for soft tissue to bone fixation in the elbow.
* Patients 18 years or older and skeletally mature.
* Patients capable of understanding the surgeon's explanations and following his/her instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study.

Exclusion Criteria:

* Infection.
* Patient conditions including blood supply limitations, and insufficient quantity or quality of bone or soft tissue.
* Patients with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions.
* Foreign body sensitivity. Where material sensitivity is suspected, testing is to be completed prior to implantation of the device.
* Patients who have any condition that would in the judgment of the Investigator place the patient at undue risk or interfere with the study.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Off-label use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had required a soft tissue to bone fixation in the elbow with the ToggleLoc 2.9 mm Soft Tissue device according to Zimmer Biomet's Instruction for Use (IFU) and and who meet all the inclusions criteria and none of the exclusions criteria.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan ACHAKRI, Study Director — Zimmer Biomet
Locations (2):
- OrthoVirginia, Fairfax, Washington, United States
- ASEPEYO Hospital, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Suffering From Biceps Tendon Rupture: Patients in need of a ToggleLoc 2.9mm in the Elbow for biceps tendon reattachment
Period: Overall Study
Arm/Group | Patients Suffering From Biceps Tendon Rupture
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Suffering From Biceps Tendon Rupture
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: "years"] | 46.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: "cm"] — Population: As only data on height on 77 cases was available, the BMI could also only be calculated for 77 cases.
  "cm"
    number analyzed (Participants) | 77
    (all) | 177.0 (7.5)
Weight [Mean (Standard Deviation); unit: "kg"] | 91.8 (19.0)
BMI [Mean (Standard Deviation); unit: "kg/m2"] — Population: As only data on height on 77 cases was available, the BMI could also only be calculated for 77 cases.
  "kg/m2"
    number analyzed (Participants) | 77
    (all) | 29.0 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue to Bone Healing in the Elbow - Hook Test
Description: Assessment of performance by analyzing soft tissue to bone healing in the elbow. The principal investigator will clinically evaluate the study elbow to assess if soft tissue to bone healing has occurred using the Hook test.
  The Hook test is performed by hooking the finger, that is inserted laterally under the biceps tendon, under the cord-like structure spanning the antecubital fossa with the patient's elbow flexed at 90 degrees.
  Each case that a Hook test was performed on will be counted as 1 count and will be described as "1 case" if successful, meaning this case had successful soft tissue to bone healing.
Time Frame: From operation to the study completion, minimum 1 year post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device
Number analyzed (Participants) | 83
Participants | 83

2. Secondary Outcome: EuroQol Five-dimensional Health Questionnaire (EQ-5D-5L): Visual Analogue Scale (VAS)
Description: Assessment of patient-reported outcome measures (PROMs): The EuroQol fivedimensional Health Questionnaire (EQ-5D-5L) is a generic instrument. The EQ-5D-5L VAS is scored on a 0 to 100 mm scale. 0 mm represents "the worst..." and 100 mm represents "the best health you can imagine".
Time Frame: At minimum 1 year post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device
Number analyzed (Participants) | 83
score on a scale | 83.3 (14.9)

3. Secondary Outcome: EuroQol Five-dimensional Health Questionnaire (EQ-5D-5L): EQ-5D-5L Profile
Description: Assessment of patient-reported outcome measures (PROMs): The EuroQol fivedimensional Health Questionnaire (EQ-5D-5L) is a generic instrument. In the EQ-5D-5L Profile the highest score is 1 and the lowest score is -0.573; negative numbers correspond to a self-assessed health state worse than being dead.
Time Frame: At minimum 1 year post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device
Number analyzed (Participants) | 83
score on a scale | 1.0 (0.1)

4. Secondary Outcome: Oxford Elbow Score (OES)
Description: Assessment of patient-reported outcome measures (PROMs): The Oxford Elbow Score (OES) consists of 12 questionnaire items with five original response options each and is specifically designed and developed for assessing outcomes of elbow surgery. The score will be on a scale from 0 (worst) to 48 (best).
Time Frame: At minimum 1 year post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device
Number analyzed (Participants) | 83
score on a scale | 46.7 (3.2)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted up to 6.1 years after surgery, when the last follow-up was performed and patients completed the study.
Description: Adverse Events were collected in an Electronic Data Capturing system called Oracle RDC, which gathers information of the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome.
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device
All-Cause Mortality (participants affected / at risk) | 0/83
Serious Adverse Events (participants affected / at risk) | 1/83
Other Adverse Events (participants affected / at risk) | 13/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ToggleLoc 2.9 mm Soft Tissue Device (N=83)
Serious Adverse Event (SAE) (Nervous system disorders) | 1 — Amyotrophic Lateral Sclerosis (ALS)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ToggleLoc 2.9 mm Soft Tissue Device (N=83)
Adverse Events (AE) (Nervous system disorders) | 1 — Median nerve dysesthesia
Adverse Events (AE) (Nervous system disorders) | 1 — Paresthesia due to tick bite
Adverse Events (AE) (Nervous system disorders) | 2 — Paresthesia
Adverse Events (AE) (Nervous system disorders) | 1 — Medium neurapraxia
Adverse Events (AE) (Nervous system disorders) | 2 — Hypoesthesia
Adverse Events (AE) (Musculoskeletal and connective tissue disorders) | 1 — Lack of Flexion and Calcifications
Adverse Events (AE) (Musculoskeletal and connective tissue disorders) | 3 — Lack of Supination
Adverse Events (AE) (Musculoskeletal and connective tissue disorders) | 1 — Heterotopic Ossification at the repair site/forearm
Adverse Events (AE) (Skin and subcutaneous tissue disorders) | 1 — Wound problems - infection

LIMITATIONS AND CAVEATS:
A limitation to this study is its retrospective design. Due to this, no data on preoperative PROMs (Oxford Elbow Score) and patient questionnaires (EQ-5D-5L Profile/VAS) were collected and therefore, no comparison to postoperative PROMs and patient questionnaires could be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05519228/Prot_SAP_000.pdf